CLINICAL TRIAL: NCT04588129
Title: An Open Label Positron Emission Tomography (PET) Study to Evaluate Dopamine Receptor Occupancy of LB-102 Administered Orally to Healthy Subjects
Brief Title: Receptor Occupancy of LB-102 Using Positron Emission Tomography (PET) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LB Pharmaceuticals Inc. (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LB-102-002
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LB-102 50 mg, single dose Cohort 1 (Experimental): LB-102 (N-Methyl amisulpride) formulated capsule will be administered orally once daily for one day in 4 subjects.
  Interventions: Drug: LB-102
- LB-102 100 mg, single dose Cohort 2 (Experimental): LB-102 (N-Methyl amisulpride) formulated capsule will be administered orally once daily for one day in 4 subjects.
  Interventions: Drug: LB-102
- LB-102 75 mg, single dose Cohort 3 (Experimental): LB-102 (N-Methyl amisulpride) formulated capsule will be administered orally once daily for one day in 4 subjects.
  Interventions: Drug: LB-102
- LB-102 100 & 50 mg, multiple dose Cohort 4 (Experimental): LB-102 (N-Methyl amisulpride) formulated capsule will be administered orally once daily for four days in 4 subjects: 2 subjects @ 100 mg and 2 subjects @ 50 mg.
  Interventions: Drug: LB-102

INTERVENTIONS:
Drug: LB-102 — (N-Methyl amisulpride)

SUMMARY:
This is an open label study in 4 cohort of 4 healthy volunteers each designed to evaluate the dopamine receptor occupancy of LB-102 at various doses and timepoints.

DETAILED DESCRIPTION:
This is a Phase 1, open label study designed to evaluate the dopamine receptor occupancy in healthy subjects. There will be 4 cohorts consisting of 4 subjects each. Eligible subjects will receive 1 or 2 doses of LB-102 on Day 1: subjects in the final cohort will be dosed for 5 days BID (ie twice/day) on an inpatient basis. This will be an open label study. Blood samples for pharmacokinetic (PK) and safety assessments will be collected at screening, immediately pre-dose, and during/before/after PET scan. Subjects enrolled in the inpatient cohort will be monitored daily. Follow-up after discharge will consist of a phone call the evening of discharge and the next day to check on subjects. This will be an adaptive study and doses in cohorts 2-4 will be determined after PET data from Cohort 1 are obtained.

ELIGIBILITY:
Inclusion Criteria:

Body Mass Index (BMI) ≥ 18 and ≤ 30 kg/m2 at screening visit. Competent to provide informed consent.

Subjects must be in good general health as determined by medical history and physical examination with no clinically significant medical findings and no history of significant medical disease (e.g., cardiovascular, pulmonary, renal, etc.) or acute condition with the past 30 days, as determined by the study investigators.

Have normal clinical laboratory test results and ECG, which are not considered to be clinically significant by the Investigator.

Exclusion Criteria:

1. Are pregnant or lactating.
2. Have a history or presence of significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological or psychological/psychiatric disorders which, in the opinion of the Investigator, increases the risk of the study drug or may confound the interpretation of study measures.
3. Clinically significant abnormal findings on physical examination or vital signs as determined by Investigator.
4. Individuals with pacemakers, aneurysm clips, shrapnel, or other restricted implanted metallic devices will be excluded from study. All subjects complete the standard MRI screening questionnaire prior to MRI.
5. History or presence of psychiatric or neurological disease or condition, as determined by the Investigator.
6. History of seizures.
7. Subject with any history or current evidence of suicidal behavior.
8. Unwilling to complete any planned study assessments.
9. Have a history of blood donation in excess of 500 mL of blood within 30 days prior to Screening.
10. Have received treatment with an investigational drug or device within 30 days prior to Screening.
11. Have a positive test for Human Immunodeficiency Virus (HIV) antibodies 1 and 2, Hepatitis B Surface Antigen (HBsAg) or Hepatitis C Virus (HCV) antibody.
12. Any subject who is known to be allergic to the study drug or any components of the study drug.
13. The subject has a fasting blood glucose ≥ 126 mg/dL or hemoglobin A1c (HbA1c) ≥ 6.5% at Screening.
14. The subject has a history of QT prolongation or dysrhythmia or a family history of prolonged QT interval or sudden death.
15. Clinically significant abnormal finding on ECG (electrocardiogram) and/or evidence of any of the following cardiac conduction abnormalities at Screening:

    1. Heart rate < 40 bpm and > 100 bpm (based on the ECG reading)
    2. QTcF interval > 450 msec for males and females
    3. PR interval ≥ 200 msec
    4. Intraventricular conduction delay with QRS duration > 120 msec
    5. Evidence of second- or third-degree atrioventricular block (AVB)
    6. Electrocardiographic evidence of complete left bundle branch block (LBBB), complete right bundle branch block (RBBB), or incomplete LBBB

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Brain Receptor Occupancy as Measured by Positron Emission Tomography | 2.5 hours post LB-102 dose
  PET scan of D2/D3 receptor occupancy using raclopride as a tracer
Brain Receptor Occupancy as Measured by Positron Emission Tomography | 7.5 hours post LB-102 dose
  PET scan of D2/D3 receptor occupancy using raclopride as a tracer
Brain Receptor Occupancy as Measured by Positron Emission Tomography | 23.5 hours post LB-102 dose
  PET scan of D2/D3 receptor occupancy using raclopride as a tracer

SECONDARY OUTCOMES:
Safety and Tolerability as Measured by Reported Adverse Events | Up to 14 days
  Measurement of clinical events as determined by medical staff reporting

CONTACTS AND LOCATIONS:
Overall Officials: Dean Wong, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Corporate Website — http://www.LBPharma.us